CLINICAL TRIAL: NCT03432533
Title: A Randomized, Multicenter, Open-label, Parallel Group Study in Postmenopausal Women With Osteoporosis to Evaluate the Noninferiority of Subject-administered Romosozumab Via Autoinjector/Pen vs Healthcare Provider-administered Romosozumab Via Prefilled Syringe
Brief Title: A Comparison of Subject-administered Romosozumab With Healthcare Provider-administered Romosozumab for Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150120; 2017-003512-40 (EudraCT Number)
Record Dates: First submitted 2018-01-30; First posted 2018-02-14 (Actual); Results first posted 2020-04-10 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Post-Menopausal Osteoporosis
Keywords: Post-Menopausal osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — romosozumab

STUDY DESIGN:
Intervention Model Description: After signing the informed consent form (ICF), subjects will undergo the following periods:
  * Screening period (35 days) to complete eligibility assessments
  * Open-label treatment period (6 months)
  * Follow-up period (3 months) During the open-label treatment period, subjects will be randomized to receive romosozumab either via HCP administration with PFS or via self-administration withAI/Pen.
  During the follow-up period, subjects will be followed for an additional 3 months to ensure appropriate follow-up for anti-romosozumab antibody formation and adverse events.
  The primary analysis will be performed after all subjects have had the opportunity to complete the Month 6 visit. The final analysis will be performed after all subjects have had the opportunity to complete the Month 9 visit.
Masking Description: This is an open-label study; blinding procedures are not applicable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Romosozumab 210 mg QM: PFS (Active Comparator): During the open-label treatment period, participants receive 210 mg romosozumab SC QM by HCP administration with PFS.
  Interventions: Drug: romosozumab HCP administration with PFS
- Romosozumab 210 mg QM: AI/Pen (Active Comparator): During the open-label treatment period, participants receive 210 mg romosozumab SC QM by self-administration with AI/pen.
  Interventions: Device: romosozumab self-administration with AI/Pen

INTERVENTIONS:
Drug: romosozumab HCP administration with PFS — 210 mg romosozumab SC QM by HCP administration with 2 PFS
  Other Names: Evenity; AMG785
  Arms: Romosozumab 210 mg QM: PFS
Device: romosozumab self-administration with AI/Pen — 210 mg romosozumab SC QM by self-administration with 2 AI/Pens
  Other Names: Evenity; AMG785
  Arms: Romosozumab 210 mg QM: AI/Pen

SUMMARY:
To evaluate the noninferiority of a 6-month treatment with 210 mg romosozumab at 90 mg/mL administered subcutaneously (SC) once a month (QM) in postmenopausal women with osteoporosis either by healthcare provider (HCP) administration with prefilled syringe (PFS) or by subject self-administration with autoinjector/pen (AI/Pen)

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent/assent prior to initiation of any studyspecific activities/procedures, or subject's legally acceptable representative has provided informed consent prior to any study-specific activities/procedures being initiated when the subject has any kind of condition that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent.
* Postmenopausal female (postmenopausal status is defined as no vaginal bleeding or spotting for 12 consecutive months prior to screening)

  -≥ 55 to ≤ 90 years of age at the time of informed consent
* Ambulatory
* BMD T-score ≤ -2.50 at the lumbar spine, total hip, or femoral neck, as assessed by the central imaging vendor at the time of screening, based on DXA scans -Subject has at least 2 vertebrae in the L1-L4 region evaluable by DXA, as assessed by the principal investigator or designee
* Subject has at least 1 hip evaluable by DXA, as assessed by the principal investigator or designee
* Subject has history of fragility (ie, osteoporosis-related fracture) or subject meets at least 2 of the following clinical risk factors for fracture

  * ≥ 70 years of age at the time of informed consent
  * BMD T-score ≤ -3.00 at the lumbar spine, total hip, or femoral neck, as assessed by the central imaging vendor at the time of screening, based on DXA scans
  * current smoker
  * consumption of ≥ 3 glasses of alcohol a day
  * parental history of fragility (ie, osteoporosis-related) fracture
  * body weight ≤ 125 pounds/56 kilogram
* Ability to follow and understand instructions and the ability to self-inject, per investigator judgement

Exclusion Criteria:

* History of osteonecrosis of the jaw and/or atypical femoral fracture
* History of metabolic or bone disease (except osteoporosis) that may interfere with the interpretation of the results, such as sclerosteosis, Paget's disease, rheumatoid arthritis, osteomalacia, osteogenesis imperfecta, osteopetrosis, ankylosing spondylitis, Cushing's disease, hyperprolactinemia, and malabsorption syndrome
* Subject with reported history of hearing loss associated with cranial nerve VIII compression due to excessive bone growth (eg, as seen in conditions such as Paget's disease, sclerosteosis and osteopetrosis)
* Vitamin D insufficiency [defined as serum 25 (OH) vitamin D levels < 20 ng/mL], as determined by the central laboratory. Vitamin D repletion will be permitted a nd subjects may be rescreened
* Current hyperthyroidism (unless well controlled on stable antithyroid therapy) by subject report or by chart review, per principal investigator evaluation
* Current clinical hypothyroidism (unless well controlled on stable thyroid replacement therapy) by subject report or by chart review, per principal investigator evaluation normal range, per subject medical history. Uncontrolled hyperparathyroidism is defined as: parathyroid hormone (PTH) outside the normal range in subjects with concurrent hypercalcemia; or PTH values > 20% above the upper limit of normal (ULN) in normocalcemic subjects.
* Current hyper- or hypocalcemia, defined as albumin-adjusted serum calcium outside the normal range, as assessed by the central laboratory. Serum calcium levels may be retested once in case of an elevated serum calcium level within 1.1x the ULN as assessed by the central laboratory

Ages: 55 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2020-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- United States (33):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Chandler, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Cypress, California
  - Research Site, Fullerton, California
  - Research Site, Glendale, California
  - Research Site, Laguna Hills, California
  - Research Site, Santa Maria, California
  - Research Site, Tustin, California
  - Research Site, Denver, Colorado
  - Research Site, Golden, Colorado
  - Research Site, Delray Beach, Florida
  - Research Site, South Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Bridgeton, Missouri
  - Research Site, Springfield, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, Great Neck, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Spartanburg, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Chesapeake, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Renton, Washington
  - Research Site, Franklin, Wisconsin
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Świdnik
  - Research Site, Warsaw
- United Kingdom (7):
  - Research Site, Chorley
  - Research Site, Edinburgh
  - Research Site, Liverpool
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Romford

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 36 centers in Poland, United Kingdom, and United States.
Pre-assignment Details: Participants were randomized in a 1:1 ratio.
Groups:
- Romosozumab 210 mg QM: PFS: During the open-label treatment period, participants received 210 mg romosozumab subcutaneously (SC) once a month (QM) by health care provider (HCP) administration with pre-filled syringe (PFS).
- Romosozumab 210 mg QM: AI/Pen: During the open-label treatment period, participants received 210 mg romosozumab SC QM by self-administration with autoinjector (AI)/pen.
Period: Overall Study
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Started | 141 | 142
Completed 6-Month Treatment Period | 136 | 137
Completed (Completed 9-Month Study Period) | 126 | 131
Not Completed | 15 | 11
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Romosozumab 210 mg QM: PFS: During the open-label treatment period, participants received 210 mg romosozumab SC QM by HCP administration with PFS.
- Romosozumab 210 mg QM: AI/Pen: During the open-label treatment period, participants received 210 mg romosozumab SC QM by self-administration with AI/pen.
- Total: Total of all reporting groups
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen | Total
Number analyzed (Participants) | 141 | 142 | 283
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (7.1) | 69.5 (8.4) | 69.9 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 142 | 283
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 138 | 141 | 279
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 139 | 140 | 279
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Lumbar Spine Bone Mineral Density (BMD) T-Score [Mean (Standard Deviation); unit: T-score] — The T-score is the BMD at the site when compared to that of a healthy thirty-year-old of the same sex. Lower scores (more negative) mean lower bone density. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5, meaning below-normal bone density without full osteoporosis; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.69 (1.03) | -2.85 (1.00) | -2.77 (1.02)
Total Hip BMD T-Score [Mean (Standard Deviation); unit: T-score] — The T-score is the BMD at the site when compared to that of a healthy thirty-year-old of the same sex. Lower scores (more negative) mean lower bone density. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5, meaning below-normal bone density without full osteoporosis; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.29 (0.73) | -2.30 (0.77) | -2.29 (0.75)
Femoral Neck BMD T-Score [Mean (Standard Deviation); unit: T-score] — The T-score is the BMD at the site when compared to that of a healthy thirty-year-old of the same sex. Lower scores (more negative) mean lower bone density. Normal is a T-score of -1.0 or higher; Osteopenia is defined as between -1.0 and -2.5, meaning below-normal bone density without full osteoporosis; Osteoporosis is defined as -2.5 or lower, meaning a bone density that is two and a half standard deviations below the mean of a thirty-year-old man/woman.
  T-score | -2.54 (0.63) | -2.49 (0.65) | -2.52 (0.64)
Participants With Pre-Existing Anti-Romosozumab Antibodies [Count of Participants; unit: Participants] — Number of participants with pre-existing antibodies, including those who were binding antibody positive and those who were neutralizing antibody positive at or before baseline (BL). Population: Participants with an assessment at baseline.
  Participants
    Binding Antibody Positive at or Before BL: number analyzed (Participants) | 139 | 141 | 280
    Binding Antibody Positive at or Before BL | 3 | 0 | 3
    Neutralizing Antibody Positive at or Before BL: number analyzed (Participants) | 139 | 141 | 280
    Neutralizing Antibody Positive at or Before BL | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine BMD at Month 6
Description: Percent change from baseline in BMD at the lumbar spine as measured by dual-energy x-ray absorptiometry (DXA).
Time Frame: Baseline, Month 6
Population: Primary Analysis Population: participants with lumbar spine BMD values at baseline and >=1 postbaseline visit at Month 6.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Number analyzed (Participants) | 135 | 134
percent change | 9.2 (0.4) | 9.0 (0.5)
Statistical Analysis 1: Comparison: Romosozumab 210 mg QM: PFS vs Romosozumab 210 mg QM: AI/Pen; Test type: Non-Inferiority — Conclusions for the primary efficacy hypothesis of efficacy of self-administration of romosozumab by AI/Pen compared with HCP-administered romosozumab by PFS at lumbar spine BMD at Month 6 was made using a 1-sided test with type 1 error rate of 0.025 and noninferiority margin of -2.0%; p = 0.84, ANCOVA; LS Mean Difference = -0.1, 95% CI 2-sided [-1.3 to 1.0], Standard Error of Mean 0.6

2. Secondary Outcome: Percent Change From Baseline in Total Hip BMD at Month 6
Description: Percent change from baseline in BMD for total hip as measured by DXA.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Number analyzed (Participants) | 135 | 134
percent change | 3.7 (0.6) | 3.6 (0.3)

3. Secondary Outcome: Percent Change From Baseline in Femoral Neck BMD at Month 6
Description: Percent change from baseline in BMD at femoral neck as measured by DXA.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Number analyzed (Participants) | 135 | 134
percent change | 3.4 (0.7) | 3.6 (0.5)

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Device-Related AEs, Discontinuations Due to AEs, and Deaths
Description: AE: any untoward medical occurrence irrespective of a causal relationship with the study treatment. SAE: any untoward medical occurrence that meets at least 1 of the following criteria: results in death; is immediately life-threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important serious event. Adverse device effect: any AE related to the use of a combination product or medical device. TEAEs are those AEs occurring after first dose of study drug.
Time Frame: up to Month 9 (-7/+3 days)
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug
Measure: Number; unit: participants
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Number analyzed (Participants) | 141 | 142
participants
  TEAEs: All | 94 | 96
  TEAEs: SAEs | 7 | 4
  TEAEs: Leading to Study Drug Discontinuation (DC) | 7 | 15
  TEAEs: Fatal | 0 | 0
  Treatment-Related (TR) TEAEs: All | 38 | 59
  TR TEAEs: SAEs | 0 | 0
  TR TEAEs: Leading to Study Drug DC | 6 | 10
  TR TEAEs: Fatal | 0 | 0
  Device-Related (DR) TEAEs: All | 18 | 30
  DR TEAEs: SAEs | 0 | 0
  DR TEAEs: Leading to Study Drug DC | 0 | 5
  DR TEAEs: Fatal | 0 | 0

5. Secondary Outcome: Number of Participants Developing Anti-Romosozumab Antibodies
Description: Participants with a negative or no result at baseline (BL) developing anti-romosozumab antibodies postbaseline, including those who were binding antibody-positive or neutralizing antibody-positive postbaseline. 'Transient' positive results are those with a negative result at the participant's last time point tested within the study period.
Time Frame: up to Month 9 (-7/+3 days)
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug as well as baseline and postbaseline antibody results.
Measure: Count of Participants; unit: Participants
Arm/Group | Romosozumab 210 mg QM: PFS | Romosozumab 210 mg QM: AI/Pen
Number analyzed (Participants) | 139 | 142
Participants
  Binding Antibody Positive Post-BL | 21 | 22
  Transient Binding Antibody Positive Post-BL | 6 | 3
  Neutralizing Antibody Positive Post-BL | 5 | 4
  Transient Neutralizing Antibody Positive Post-BL | 0 | 2

ADVERSE EVENTS:
Time Frame: up to Month 9 (-7/+3 days)
Description: All-cause mortality is reported for all participants enrolled/randomized in the study. Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug.
Groups:
- Romosozumab 210 mg SC QM by PFS: During the open-label treatment period, participants received 210 mg romosozumab SC, QM by HCP administration with PFS.
- Romosozumab 210 mg SC QM by AI/Pen: During the open-label treatment period, participants received 210 mg romosozumab SC QM by self-administration with AI/pen.
Arm/Group | Romosozumab 210 mg SC QM by PFS | Romosozumab 210 mg SC QM by AI/Pen
All-Cause Mortality (participants affected / at risk) | 0/141 | 0/142
Serious Adverse Events (participants affected / at risk) | 7/141 | 4/142
Other Adverse Events (participants affected / at risk) | 48/141 | 64/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romosozumab 210 mg SC QM by PFS (N=141) | Romosozumab 210 mg SC QM by AI/Pen (N=142)
Myocardial infarction (Cardiac disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romosozumab 210 mg SC QM by PFS (N=141) | Romosozumab 210 mg SC QM by AI/Pen (N=142)
Injection site erythema (General disorders) | 25 | 35
Injection site pain (General disorders) | 14 | 21
Injection site swelling (General disorders) | 11 | 23
Nasopharyngitis (Infections and infestations) | 15 | 10
Upper respiratory tract infection (Infections and infestations) | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 9
Headache (Nervous system disorders) | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03432533/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03432533/SAP_001.pdf